CLINICAL TRIAL: NCT03871816
Title: Biomarker Study to Determine Frequency of DNA-repair Defects in Men With Metastatic Prostate Cancer
Brief Title: A Study to Determine Frequency of DNA-repair Defects in Men With Metastatic Prostate Cancer
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR108591; 64091742PCR0002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-03-11; First posted 2019-03-12 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Metastatic Prostate Cancer: Participants with metastatic prostate Cancer (PC) will be evaluated for the prevalence of DNA-repair gene defects (DRDs) and will be assessed for biomarker eligibility status for niraparib interventional studies. Participants will be consented to saliva, blood, and/or archival tumor tissue testing for the presence or absence of DNA-repair gene defects.
  Interventions: Other: Saliva, Blood, or and/or Archival Tumor Tissue Collection and Analysis

INTERVENTIONS:
Other: Saliva, Blood, or and/or Archival Tumor Tissue Collection and Analysis — Saliva, blood, and/or archival tumor tissue will be collected from the participants with metastatic PC for genomic testing to confirm DRD status.

SUMMARY:
The purpose of this study is to evaluate the prevalence of 4 or more DNA-repair gene defects in a population of men with metastatic Prostate Cancer (PC) and to use the reported DNA-repair gene defects to assess biomarker eligibility for niraparib interventional studies.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic (Stage IV) prostate cancer (PC), confirmed by either biopsy of a metastatic tumor site or history of localized disease supported by metastatic disease on imaging studies (that is [i.e.], clearly noted in hospital/clinical records)
* Signed Informed consent form (ICF)
* No condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant (for example [e.g.], compromise the well-being) or that could prevent, limit, or confound the protocol-specified assessments
* Willing to provide a saliva, blood, and/or archival tumor tissue sample for genomic analysis
* No prior poly (adenosine diphosphate [ADP]-ribose) polymerase inhibitor (PARPi) for the treatment of prostate cancer
* No prior DNA-repair gene defect test results from a Janssen sponsored interventional trial

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population consists of male participants diagnosed with metastatic prostate cancer who will be evaluated for the prevalence for DNA-repair gene defects.
Sampling Method: Probability Sample
Enrollment: 14532 (Actual)
Dates: Start 2019-04-22 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-11-22 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with 4 or more DNA-repair Gene Defects with Metastatic Prostate Cancer as an Estimate for Prevalence | Approximately 2.4 years
  Percentage of participants with 4 or more Deoxyribonucleic acid (DNA)-repair gene defects with metastatic Prostate Cancer (PC) as an estimate for prevalence will be assessed. A saliva, blood, and/or archival tumor tissue sample will be collected for genomic testing to confirm DNA-repair gene defect (DRD) status.
Percentage of Participants who Meet Biomarker Eligibility Criteria for Other Niraparib Interventional Studies | Approximately 2.4 years
  Percentage of participants who meet biomarker eligibility criteria for other niraparib interventional studies will be assessed.

SECONDARY OUTCOMES:
Percentage of Participants with 4 or more DNA-repair Gene Defects with Metastatic Castration-Resistant Prostate Cancer (mCRPC) and with Metastatic Hormone Sensitive PC (HSPC) as an Estimate for Prevalence | Approximately 2.4 years
  Percentage of participants with 4 or more DRDs with mCRPC and HSPC as an estimate for prevalence will be assessed. A saliva, blood, and/or archival tumor tissue sample will be collected for genomic testing to confirm DRD status.
Percentage of Participants with 1 or more DNA-repair gene defects with Metastatic Prostate Cancer as an Estimate for Prevalence | Approximately 2.4 years
  Percentage of participants with 1 or more DRDs with metastatic PC as an estimate for prevalence will be assessed. Saliva, blood, and/or archival tumor tissue sample will be collected for genomic testing to confirm DRD status.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (338):
- United States (93):
  - Urology Centers Of Alabama, Homewood, Alabama
  - Southern Cancer Center, PC, Mobile, Alabama
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Mayo Clinic, Phoenix, Arizona
  - Urological Associates of Southern Arizona, P.C., Tucson, Arizona
  - Yuma Regional Medical Center, Yuma, Arizona
  - Arkansas Urology, Little Rock, Arkansas
  - MemorialCare Research Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Kaiser Permanente, Riverside, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Sansum Clinic Pharm, Santa Barbara, California
  - Rocky Mountain Cancer Centers, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Foothills Urology - Golden Off, Golden, Colorado
  - Eastern Connecticut Hematology & Oncology Assoc., Norwich, Connecticut
  - Advanced Urology Institute, Daytona Beach, Florida
  - Holy Cross Hospital - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Cancer Specialists of North Florida, Jacksonville, Florida
  - Miami Cancer Institute at Baptist Health / Baptist Health Medical Group, Miami, Florida
  - Ocala Oncology Center, Ocala, Florida
  - Woodlands Medical Specialists, PA, Pensacola, Florida
  - University Cancer & Blood Center, LLC, Athens, Georgia
  - Hawaii Cancer Care, Honolulu, Hawaii
  - Affiliated Oncologists, LLC, Chicago Ridge, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - First Urology, Jeffersonville, Indiana
  - Beacon Medical Group Clinical Research, South Bend, Indiana
  - Norton Healthcare, Louisville, Kentucky
  - Pontchartrain Cancer Center, Covington, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Maryland Oncology Hematology, PA, Columbia, Maryland
  - Frederick Health Hospital - James M Stockman Cancer Institute, Frederick, Maryland
  - Chesapeake Urology Associates, Towson, Maryland
  - Beth Israel Deaconess Hospital Plymouth, Jordan Club Cancer Center, Plymouth, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Edward W Sparrow Hospital, Lansing, Michigan
  - Michigan Institute of Urology, Troy, Michigan
  - Minnesota Oncology Hematology, P.A., Minneapolis, Minnesota
  - Central Care Cancer Center, Bolivar, Missouri
  - Mosaic Life Care, Saint Joseph, Missouri
  - Adult Pediatric Urology & Urogynecology, P.C, Omaha, Nebraska
  - GU Research Network, Omaha, Nebraska
  - Nebraska Cancer Specialists, Omaha, Nebraska
  - New York Oncology Hematology, Albany, New York
  - Tisch Cancer Institution, New York, New York
  - Associated Medical Professionals, Syracuse, New York
  - Upstate Cancer Center, Syracuse, New York
  - Montefiore Medical Center, The Bronx, New York
  - Southeastern Medical Oncology Center, Goldsboro, North Carolina
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Willamette Valley Cancer Institute and Research Center, Eugene, Oregon
  - Northwest Cancer Specialists PC, Portland, Oregon
  - Oregon Oncology Specialists, Salem, Oregon
  - Oregon Urology Institute, Springfield, Oregon
  - Centers for Advanced Urology LLC d b a MidLantic Urology, Bala-Cynwyd, Pennsylvania
  - Gettysburg Cancer Center, Gettysburg, Pennsylvania
  - Consultants in Medical Oncology and Hematology, P.C. - Abington, Horsham, Pennsylvania
  - Lancaster Urology, Lancaster, Pennsylvania
  - University of Pittsburgh Medical Center (UPMC), Pittsburgh, Pennsylvania
  - Prisma Health, Greenville, South Carolina
  - Atlantic Urology Clinics, Myrtle Beach, South Carolina
  - Texas Onc., Abilene, Texas
  - Texas Oncology-Amarillo, Amarillo, Texas
  - Texas Oncology-Austin, Austin, Texas
  - Texas Oncology-Beaumont, Mamie McFaddin Ward Cancer Center, Beaumont, Texas
  - Methodist Dallas Medical Center, Dallas, Texas
  - Texas Oncology-Denton South, Denton, Texas
  - Texas Oncology, P.A. - Flower Mound, Flower Mound, Texas
  - Texas Oncology-Fort Worth Cancer Center, Fort Worth, Texas
  - Texas Oncology-Memorial City, Houston, Texas
  - Houston Metro Urology, Houston, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology - Willowbrook, Houston, Texas
  - Texas Oncology P.A., Longview, Texas
  - Texas Oncology P.A., McAllen, Texas
  - Texas Oncology-Mesquite, Mesquite, Texas
  - Texas Oncology-Midland Allison Cancer Center, Midland, Texas
  - Texas Oncology, P.A. - Paris, Paris, Texas
  - Texas Oncology P A, Plano, Texas
  - Texas Oncology P.A., Plano, Texas
  - University of Texas at San Antonio, San Antonio, Texas
  - Texas Oncology -Waco, Waco, Texas
  - Texas Oncology Deke Slayton Cancer Center, Webster, Texas
  - Texas Oncology P.A., Wichita Falls, Texas
  - University of Virginia, Charlottesville, Virginia
  - INOVA, Fairfax, Virginia
  - Virginia Cancer Specialists, Leesburg, Virginia
  - Virginia Oncology Asc, Norfolk, Virginia
  - Urology of Virginia, PLCC, Virginia Beach, Virginia
  - Northwest Medical Specialists, Tacoma, Washington
  - Building Oncology Research, Janesville, Wisconsin
  - University of Wisconsin Carbone Cancer Center, Madison, Wisconsin
- Argentina (15):
  - Hospital Aleman, Buenos Aires
  - Sociedade Beneficente de Senhoras - Hospital Sírio Libanês, Buenos Aires
  - Centro Oncológico Korben, Buenos Aires
  - CEMIC Saavedra, Buenos Aires
  - CINME - Centro de Investigaciones Metabolicas, Caba
  - Centro de Urologia (CDU), Ciudad Automoma Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma de
  - Clínica Adventista Belgrano, Ciudad de Buenos Aires
  - Cemaic - Centro Privado de Especialidades Medicas Ambulatorias e Investigacion Clinica, Córdoba
  - Centro Urologico Profesor Bengio, Córdoba
  - Hospital Privado - Centro Medico de Cordoba, Córdoba
  - Hospital Privado de Comunidad, Mar del Plata
  - Centro de Investigacion Pergamino SA, Pergamino
  - Sanatorio Parque, Rosario
  - ARS Médica, San Salvador de Jujuy
- Australia (13):
  - Pindara Private Hospital, Benowa
  - Sunshine Coast University Hospital, Birtinya
  - Chris O'Brien Lifehouse, Camperdown
  - St Vincent's hospital, Darlinghurst
  - Border Medical Oncology, East Albury
  - Royal Hobart Hospital, Hobart
  - Ashford Cancer Centre, Kurralta Park
  - Liverpool Hospital, Liverpool
  - Macquarie University Hospital, Macquarie University
  - Peter MacCallum Cancer Centre, Melbourne
  - Fiona Stanley Hospital, Murdoch
  - Prince Of Wales Hospital, Randwick
  - Sydney Adventist Hospital, Wahroonga
- Belarus (8):
  - Bobruisk Interregional Oncological Dispensary, Babruysk
  - Brest Regional Oncology Dispensary, Brest
  - Grodno University Hospital, Grodno
  - Gomel Regional Clinical Oncology Dispensary, Homyel
  - State Institution N.N. Alexandrov Republican Scientific and, Lesnoy
  - Minsk city Clinical Oncological Dispensary, Minsk
  - Mogilev Regional Hospital, Mogilev
  - Vitebsk Regional Clinical Hospital, Vitebsk
- Belgium (4):
  - Clinique Notre Dame de Grâce, Charleroi
  - Jolimont, Haine-Saint-Paul, La Louviere
  - Clinique Saint Pierre, Ottignies
  - Algemeen Ziekenhuis Delta, Roeselare
- Brazil (34):
  - Fundacao Pio XII, Barretos
  - Cetus Oncologia, Belo Horizonte
  - PERSONAL - Oncologia de Precisão e Personalizada, Belo Horizonte
  - Sociedade Beneficente de Senhoras - Hospital Sirio Libanes HSL Unidade Brasilia, Brasília
  - CIONC - Centro Integrado de Oncologia de Curitiba, Curitiba
  - Liga Paranaense de Combate ao Cancer, Curitiba
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina - CEPEN, Florianópolis
  - Suporte Nutricional e Quimioterapia Ltda-Pronutrir, Fortaleza
  - Associacao de Combate ao Cancer em Goias - Hospital de Cancer Araujo Jorge, Goiânia
  - Oncosite - Centro de Pesquisa Clínica em Oncologia Ltda, Ijuí
  - Fundação São Francisco Xavier, Ipatinga
  - Clínica de Neoplasias Litoral Ltda., Itajaí
  - Instituto Joinvilense de Hematologia e Oncologia Ltda-Centro de Hematologia e Oncologia, Joinville
  - Medradius Clinica de Medicina Nuclear e Radiologia de Maceio Ltda., Maceió
  - Liga Norte Riograndense Contra O Cancer, Natal
  - Irmandade Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Hospital Ernesto Dornelles, Porto Alegre
  - MultiHemo Servicos Medicos S.A, Recife
  - Universidade do Estado do Rio de Janeiro - UERJ, Rio de Janeiro
  - Oncoclínicas Rio de Janeiro S.A., Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Nucleo de Oncologia da Bahia, Salvador
  - Hospital Sao Rafael, Salvador
  - CEPHO - Centro de Estudos e Pesquisa de Hematologia e Oncologia, Santo André
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo
  - Irmandade Santa Casa de Misericordia de Sao Paulo, São Paulo
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Fundacao Faculdade de Medicina - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo
  - Fundacao Antonio Prudente - A.C. Camargo Cancer Center, São Paulo
  - Núcleo de Pesquisa São Camilo, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual - IAMSPE, São Paulo
  - IOS - Instituto de Oncologia de Sorocaba Dr. Gilson Delgado, Sorocaba
  - Instituto do Cancer De Tres Lagoas, Três Lagoas
- Bulgaria (4):
  - MHAT Deva Maria, Burgas
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - District Oncology Dispensary with In-Patient Stationary - Plovdiv, Plovdiv
  - Comprehensive Cancer Center, Vratsa
- Canada (8):
  - Southern Alberta Institute of Urology / Prostate Cancer Centre, Calgary, Alberta
  - British Columbia Cancer Agency (BCCA) - Vancouver Centre, Vancouver, British Columbia
  - British Columbia Cancer Agency - Vancouver Island Centre, Victoria, British Columbia
  - McMaster Institute of Urology, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario (Kingston Regional Cancer Centre), Kingston, Ontario
  - University Health Network (UHN) Princess Margaret Cancer Centre, Toronto, Ontario
  - Centre de Recherche du CHUM, Montreal, Quebec
  - Centre hospitalier universitaire de Québec (CHUQ), L'Hotel-Dieu de Quebéc, Québec, Quebec
- Denmark (2):
  - Copenhagen University Hospital, Copenhagen
  - Næstved Hospital, Næstved
- France (17):
  - Institut Sainte Catherine, Avignon
  - Centre Hospitalier Regional Universitaire Besancon, Besançon
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Oscar Lambret, Lille
  - Centre Leon Bérard, Lyon
  - Polyclinique de Gentilly, Nancy
  - Centre Antoine Lacassagne, Nice
  - Hopital Europeen Georges-Pompidou, Paris
  - Institut de Cancérologie de l'Ouest (ICO), Saint-Herblain
  - HIA Begin, Saint-Mandé
  - Institut de Cancérologie de Loire, Saint-Priest-en-Jarez
  - Clinique Sainte Anne, Strasbourg
  - Hôpitaux Universitaire de Strasbourg -CHU, Strasbourg
  - Hopital Foch, Suresnes
  - CHRU de Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Germany (8):
  - Urologisches Zentrum Bonn, Bonn
  - Urologie im Schlosscarree Schreier/Eichler/Junius - Germany, Braunschweig
  - Zeisigwaldkliniken Bethanien Chemnitz, Chemnitz
  - Urologische Gemeinschaftspraxis Böhm/Linne - Germany, Dresden
  - uro Eimsbüttel - Gemeinschaftspraxis Bath/Weinzierl, Hamburg
  - Klinikum Region Hannover Klinikum Siloah, Hanover
  - Matthias Schulze - Germany, Markkleeberg
  - CUROS - Uberörtliche urologische Gemeinschaftspraxis, Wesseling
- Israel (5):
  - Soroka Hospital, Beersheba
  - Rambam Hospital, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Asaf Harofe Medical Center, Zrifin
- Italy (15):
  - Ospedale Cardinal Massaia, Asti
  - Ospedale Sacro Cuore Di Gesu, Benevento
  - Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Ospedale di Bolzano, Bolzano
  - oncologia medica - Oncology, Brindisi
  - Azienda Ulss 6 Euganea- Ospedale Di Camposampiero, Camposampiero
  - Ospedale Di Carrara, Carrara
  - AORN Sant'anna e San Sebastiano, Caserta
  - ASST -Ospedale Maggiore di Crema, Crema
  - Azienda ULSS 3 Serenissima, presidio di Mirano, Mirano
  - PP.OO. di Piombino e Portoferraio Azienda USL Toscana nord ovest, Piombino
  - Ospedale degli Infermi, Ponderano
  - Ospedale del Mare ASL Napoli 1 centro, Ponticelli
  - Azienda ULSS5 Polesana di Rovigo - Ospedale Santa Maria della Misericordia, Rovigo
  - PO Ospedale S.Anna, ASST Lariana, San Fermo della Battaglia
- Malaysia (4):
  - Hospital Pulau Pinang, George Town
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Sarawak General Hospital, Kuching
- Netherlands (3):
  - Renier de Graaf, Delft
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
- Poland (9):
  - Centrum Onkologii im. Prof. F. Lukaszczyka, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Szpitale Pomorskie Sp. z o.o., Gdynia
  - Przychodnia Lekarska KOMED Roman Karaszewski, Konin
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Lodzi, Lodz
  - Urologica Praktyka Lekarska Adam Marcheluk, Siedlce
  - Narodowy Instytut Onkologii im Marii Sklodowskiej Curie Panstwowy Instytut Badawczy, Warsaw
  - Szpital Grochowski im. dr med. Rafała Masztaka Sp. z o.o., Warsaw
  - Specjalistyczna przychodnia lekarska POLIMED, Wroclaw
- Russia (13):
  - Altai Regional Oncology Dispensary, Barnaul
  - Chelyabinsk Regional Clinical Center Of Oncology And Nuclear Medicine, Chelyabinsk
  - Ivanovo Regional Oncology Dispensary, Ivanovo
  - Russian Scientific Center of Roentgenoradiology, Moscow
  - Moscow City Clinical Hospital # 62, Moscow
  - Hertzen Oncology Research Institute, Moscow
  - Privolzhsky District Medical Centre, Nizhny Novgorod
  - Clinical Oncology Dispensary, Omsk
  - Pyatigorsk Interdistrict Oncology Dispensary, Pyatigorsk
  - Leningrad Regional Oncology Dispensary, Saint Petersburg
  - Republican Oncology Dispensary, Saransk
  - Multifunctional clinical medical center 'Medical city', Tyumen
  - Bashkir State Medical University, Ufa
- South Korea (14):
  - Pusan National University Hospital, Busan
  - Kyungpook National University Chilgok Hospital, Daegu
  - Keimyung University Dongsan Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - National Cancer Center, Goyang-si
  - Chonnam National University Hospital, Gwangju
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul
- Spain (25):
  - Hosp. Univ. A Coruna, A Coruña
  - Hosp. de La Santa Creu I Sant Pau, Barcelona
  - Hosp. Clinic de Barcelona, Barcelona
  - Hosp. Gral. Univ. de Castellon, Castellon
  - Institut Català D'Oncologia Girona, Girona
  - Hosp. Univ. de Jaen, Jaén
  - Hosp. de Jerez de La Frontera, Jerez de la Frontera
  - Hosp. Univ. Arnau de Vilanova de Lleida, Lleida
  - Hosp. Univ. de La Princesa, Madrid
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Hm Monteprincipe, Madrid
  - Hosp. Univ. Del Henares, Madrid
  - Hosp. Virgen de La Victoria, Málaga
  - Complexo Hosp. Univ. de Ourense, Ourense
  - Hosp. Univ. Infanta Cristina, Parla, Madrid
  - Hosp. Puerto Real, Puerto Real, Cádiz
  - Corporacio Sanitari Parc Tauli, Sabadell
  - Hosp. Univ. Marques de Valdecilla, Santander
  - Hosp. Virgen Del Rocio, Seville
  - Hosp. de Sant Pau I Santa Tecla, Tarragona
  - Hosp. de Terrassa, Terrassa
  - Hosp. Clinico Univ. de Valencia, Valencia
- Sweden (2):
  - Skanes universitetssjukhus, Malmo
  - Södersjukhuset, Stockholm
- Taiwan (10):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Tungs' Taichung MetroHarbor Hospital, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center - Yong Kang, Tainan
  - National Taiwan University Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Thailand (3):
  - Ramathibodi Hospital, Bangkok
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (11):
  - Dr.Abdurrahman Yurtaslan Oncology Training and Research Hospital, Ankara
  - Memorial Ankara Hastanesi, Ankara
  - Ankara Bilkent City Hospital, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Bursa Yuksek lhtisas EAH Medikal Onkoloji Klinigi, Bursa
  - Trakya University Medical Faculty, Edirne
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Istanbul Universitesi Cerrahpasa Tip Fakultesi Ic Hastaliklari Anabilim Dali Medikal Onkoloji Bd, Istanbul
  - T.C. Saglik Bakanlıgi Goztepe Prof. Dr. Suleyman Yalcın Sehir Hastanesi, Istanbul
  - Izmir Medical Park Hospital, Izmir
  - Sakarya University Training and Research Hospital, Sakarya
- Ukraine (15):
  - Communal Nonprofit Enterprise 'Cherkasy Regional Oncology Dispensary Of Cherkasy Regional Council', Cherkasy
  - Ce 'Dnipropetrovsk Regional Clinical Hospital N.A. Mechnikov' of Dnipropetrovsk Rc, Dnipo
  - Municipal Institution 'Clinical Oncology Dispensary' Under Dnipropetrovsk Regional Council, Dnipro
  - Ivano-Frankivsk Regional Clinical Hospital, Ivano-Frankivsk
  - Communal Institution 'City hospital №7 of Kamianske' of Dnepropetrov'sk Regional Council, Kamianske
  - Municipal non-profit enterprise 'Regional Center of Oncology', Khakhiv
  - Regional Medical Clinical Center for Urology and Nephrology named after V.I. Shapoval, Kharkiv
  - Khmelnitckiy regional hospital, Khmelnytsky
  - Communal Nonprofit Enterprise 'Regional Clinical Oncology Center of Kirovohrad Regional Council', Kropyvnytskyi
  - National Cancer Institute, Kyiv
  - State Institution Institute of Urology NAMS of Ukraine based on Kyiv City Clinical Oncology Center, Kyiv
  - Lviv Clinical Regional Hospital, Lviv
  - ME 'Poltava Regional Clinical Hospital n.a. M.V. Sklifosovsky of the Poltava Regional Council', Poltava
  - Municipal Oncology Centre of Uzhgorod Central Municipal Clinical Hospitlal, Uzhhorod
  - Communal Institution 'Regional Oncology Dispensary' of Zhytomyr Region Council, Zhytomyr
- United Kingdom (3):
  - Royal Blackburn Hospital, Blackburn
  - Royal Marsden Hospital, London
  - University College London Hospitals, London